CLINICAL TRIAL: NCT04530539
Title: The Effect of Melatonin and Vitamin C on COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020-68
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: vitamin c; melatonin
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Ascorbic Acid; Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental- Melatonin (Experimental): Patients will receive melatonin
  Interventions: Dietary Supplement: melatonin; Other: Symptom Survey
- Experimental- Vit C (Experimental): Patients will receive vitamin C
  Interventions: Dietary Supplement: Vitamin C; Other: Symptom Survey
- Control (Placebo Comparator): Patients will receive placebo
  Interventions: Dietary Supplement: Placebo; Other: Symptom Survey

INTERVENTIONS:
Dietary Supplement: Vitamin C — 1000mg Vitamin C, at bedtime
  Other Names: ascorbic acid
  Arms: Experimental- Vit C
Dietary Supplement: melatonin — 10mg melatonin, at bedtime
  Arms: Experimental- Melatonin
Dietary Supplement: Placebo — Placebo at bedtime
  Arms: Control
Other: Symptom Survey — Daily symptom survey to be completed by patient electronically

SUMMARY:
This is a double-blind placebo controlled trial that seeks to evaluate the impact of melatonin and vitamin C on symptoms and outcomes of patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria

* COVID-19 positive test (outpatient testing),
* Age >50 (chosen based greater risk for older patients to be vitamin deficient, age >65 not used so as not to be too restrictive in the inclusion criteria)
* Experiencing symptoms for <5 days prior to enrollment
* Able to read and write in English or Spanish
* Able to access REDCap daily
* Valid email address
* Current has a Lancaster General Health primary care physician

Exclusion Criteria

* COVID-19 test ordered pre-procedure for asymptomatic screening
* Currently taking vitamin C supplements
* Currently taking melatonin supplements
* Currently hospitalized
* Deceased
* Currently pregnant
* Currently incarcerated

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Symptom Severity | 14 days
  Symptom severity will be tracked electronically

SECONDARY OUTCOMES:
Symptom progression | 14 days
  Determine symptom course of those with moderate or severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Corey Fogleman, Principal Investigator — Penn Medicine Lancaster General Health; Corey Fogleman, MD, Principal Investigator — Physician
Locations (1):
- Lancaster General Health, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No